CLINICAL TRIAL: NCT03011034
Title: A Phase 2 Proof-of-Concept Study to Separately Evaluate the Activity of Talacotuzumab (JNJ-56022473) or Daratumumab in Transfusion-Dependent Subjects With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) Who Are Relapsed or Refractory to Erythropoiesis-Stimulating Agent (ESA) Treatment
Brief Title: Study to Separately Evaluate the Activity of Talacotuzumab (JNJ-56022473) or Daratumumab in Transfusion-Dependent Participants With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS) Who Are Relapsed or Refractory to Erythropoiesis-Stimulating Agent (ESA) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108261; 2016-003328-22 (EudraCT Number); 56022473MDS2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Talacotuzumab (Experimental): Participants will receive talacotuzumab 9 milligram per kilogram (mg/kg) intravenously (IV) on Days 1 and 15 for all cycles. Each treatment cycle is of 28 days. The talacotuzumab arm of the study is closed for enrollment.
  Interventions: Drug: Talacotuzumab
- Daratumumab (Experimental): Participants will receive daratumumab 16 mg/kg IV on Days 1, 8, 15, and 22 for Cycles 1 and 2; on Days 1 and 15 for Cycles 3 to 6; and on Day 1 for all subsequent cycles. Each treatment cycle is of 28 days.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Talacotuzumab — Talacotuzumab 9 mg/kg will be administered as an IV infusion.
  Other Names: JNJ-56022473
  Arms: Talacotuzumab
Drug: Daratumumab — Daratumumab 16 mg/kg will be administered as an IV infusion.
  Other Names: JNJ-54767414
  Arms: Daratumumab

SUMMARY:
The main purpose of the study is to evaluate the efficacy (transfusion independence [TI]) of talacotuzumab (JNJ-56022473) or daratumumab in transfusion-dependent participants with low or intermediate-1 risk Myelodysplastic Syndrome (MDS) whose disease has relapsed during treatment with or is refractory to Erythropoiesis-Stimulating Agent (ESAs).

DETAILED DESCRIPTION:
This is a multicenter, randomized (study drug assigned by chance), open-label (participants and researchers are aware of the treatment participants are receiving) study to evaluate the safety and efficacy of talacotuzumab or daratumumab. Approximately 60 participants (30 to receive talacotuzumab and 30 to receive daratumumab) will be enrolled and then assigned randomly on a 1:1 basis to receive either talacotuzumab or daratumumab. The study consists of: a Screening Phase of up to 28 days during which participant eligibility will be reviewed and approved by the sponsor prior to randomization, a Treatment Phase that will extend from the first dose on Cycle 1 Day 1 until study drug discontinuation, and a Post-treatment Follow up Phase beginning once the participant discontinues talacotuzumab or daratumumab. Study drugs will continue to be administered until disease progression, lack of response, unacceptable toxicity, withdrawal of consent, or study end. Safety will be monitored throughout the study. The talacotuzumab arm of the study is closed for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic Syndrome (MDS) according to World Health Organization (WHO) criteria confirmed by bone marrow aspirate and biopsy within 12 weeks prior to first dose. A local laboratory report from this diagnostic bone marrow aspirate and biopsy must be approved by the sponsor
* International Prognostic Scoring System (IPSS) low risk or intermediate-1 risk MDS
* Red blood cell (RBC) transfusion dependent, 1) Received at least 4 units of RBCs over any 8 consecutive weeks during the 16 weeks prior to randomization, 2) Pretransfusion Hb must have been less than or equal to (<=)9.0 gram per deciliter (g/dL)
* Adequate iron stores, defined as transferrin saturation greater than 20 percent (%) and serum ferritin greater than 400 nanogram per Milliliter (ng/mL), measured within the screening period, or adequate iron stores as demonstrated by recent (within 12 weeks prior to first dose) bone marrow examination with iron stain
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to talacotuzumab and daratumumab or their excipients
* Received any chemotherapy, immunomodulatory or immunosuppressive therapy, corticosteroids (greater than [>]30 milligram per day [mg/day] prednisone or equivalent) within 28 days prior to randomization
* Received other treatments for MDS within 28 days prior to first dose (example [eg], azacitidine, decitabine, lenalidomide, Erythropoiesis-Stimulating Agent (ESA) (8 weeks for long-acting ESAs)
* History of hematopoietic stem cell transplant
* Del(5q) karyotype unless treatment with lenalidomide has failed. Failure is defined as either: 1) having received at least 3 months of lenalidomide treatment without RBC transfusion benefit (International Working Group [IWG] 2006); 2) progression or relapse after hematologic improvement with lenalidomide (IWG 2006); 3) discontinuation of lenalidomide due to toxicity; or 4) unable to receive lenalidomide due to a contraindication. Source documentation for lenalidomide treatment failure must be verified by the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (21):
- United States (3):
  - Washington University School Of Medicine, St Louis, Missouri
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Belgium (4):
  - ZNA Stuivenberg, Antwerp
  - Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - AZ Turnhout, Turnhout
- Italy (4):
  - Azienda Opedaliero-Universitaria Policlinico Sant'orsola Malpighi di Bologna, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Pad. Marcora, Milan
  - Istituto Clinico Humanitas, Rozzano
- Netherlands (3):
  - UMCG, Groningen
  - Erasmus MC, Rotterdam
  - Haga ziekenhuis, The Hague
- Russia (3):
  - City Clinical Hospital # 40, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Saint Petersburg City Hospital #15, Saint Petersburg
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. I Politecni La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 34 enrolled participants, 33 participants received daratumumab and 1 participant received talacotuzumab.
Pre-assignment Details: Due to serious infusion-related reaction (IRR) event that occurred in first participant enrolled in talacotuzumab arm, no further participants were enrolled in this arm.
Groups:
- Talacotuzumab: Participant received a single dose of talacotuzumab 9 milligram per kilogram (mg/kg) intravenously (IV).
- Daratumumab: Participants received daratumumab 16 mg/kg IV weekly on Weeks 1 to 8 (on Days 1, 8, 15, and 22 for Cycles 1 and 2), every 2 weeks for Weeks 9 to 24 (on Days 1 and 15 for Cycles 3 to 6), and every 4 weeks thereafter (on Day 1 for all subsequent cycles). Each treatment cycle was 28 days.
Period: Overall Study
Arm/Group | Talacotuzumab | Daratumumab
Started | 1 | 33
Completed | 0 | 33
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Talacotuzumab | Daratumumab | Total
Number analyzed (Participants) | 1 | 33 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 | 71.5 (6.86) | 71.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 1 | 25 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 1 | 27 | 28
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Other | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
  White | 1 | 29 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 1 | 6 | 7
  ITALY | 0 | 3 | 3
  NETHERLANDS | 0 | 3 | 3
  RUSSIAN FEDERATION | 0 | 3 | 3
  SPAIN | 0 | 10 | 10
  UNITED STATES | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence (TI) Lasting at Least 8 Weeks
Description: Percentage of participants who achieved RBC TI lasting at least 8 weeks were reported. RBC TI was defined as absence of RBC transfusion during any consecutive 56 days (8 weeks) post randomization.
Time Frame: Up to 2 years
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 6.1 [0.7 to 20.2]

2. Secondary Outcome: Percentage of Participants Who Achieved Red Blood Cell (RBC) Transfusion Independence (TI) Lasting at Least 24 Weeks
Description: Percentage of participants who achieved RBC TI lasting at least 24 weeks were reported. RBC TI was defined as absence of RBC transfusion during any consecutive 56 days (8 weeks) post randomization.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 3.0 [0.1 to 15.8]

3. Secondary Outcome: Time to Transfusion Independence (TI)
Description: Time to transfusion independence (TI) was defined as time to the start of the TI interval. TI was defined as absence of RBC transfusion during any consecutive 56 days (8 weeks) post randomization.
Time Frame: Up to 2 years
Population: ITT population who achieved TI for at least 8 weeks. As less number of participants were evaluable for this outcome measure (OM), the results were not summarized. Hence, participant wise data is reported.
Measure: Number; unit: Weeks
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 2
Weeks
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 4
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 5
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | NA — Here, NA signifies that time to TI could not be estimated as this participant did not achieve TI. |

4. Secondary Outcome: Duration of Transfusion Independence (TI)
Description: Duration of TI was reported. TI was defined as absence of RBC transfusion during any consecutive 56 days (8 weeks) post randomization.
Time Frame: Up to 2 years
Population: as for outcome 3
Measure: Number; unit: Weeks
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 2
Weeks
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 16
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 65
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | NA — Here, NA signifies that duration of TI could not be estimated as this participant did not achieve TI. |

5. Secondary Outcome: Percentage of Participants Who Met IWG Criteria for Transfusion Reduction
Description: Percentage of participants who met IWG criteria for transfusion reduction were reported. IWG criteria for transfusion reduction: at least 4 units reduction in RBC transfusions in the best 8-week interval. The best 8-week interval was a post-baseline 8-week interval where the participant had the fewest post-baseline RBC transfusion units.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 54.5

6. Secondary Outcome: Percentage of Participants With at Least One Dose of Myeloid Growth Factors Usage
Description: Percentage of participants with Myeloid Growth Factors (MGF) usage (who had used at least 1 dose of MGF) were reported.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 9.1

7. Secondary Outcome: Percentage of Participants With Hematologic Improvement (HI) Per IWG 2006 by Investigator Assessment
Description: Percentage of participants with HI per International Working Group (IWG) 2006 by investigator assessment were reported. Response criteria per IWG 2006 for HI: Erythroid response (pretreatment, less than [<]11 gram per deciliter [g/dL]) - hemoglobin increase by greater than or equal to (>=)1.5 g/dL, relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for a Hb of <=9 g/dL pretreatment counted in the RBC transfusion response evaluation; Platelet response (pretreatment, <100*10^9/L) - absolute increase of >=30*10^9/L for participants starting with >20*10^9/L platelets. Increase from <20*10^9/L to >20*10^9/L and by at least 100 percent (%); Neutrophil response (pretreatment, <1*10^9/L) - at least 100% increase and an absolute increase >0.5*10^9/L.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants
  Erythroid Response | 0 | 9.1 [1.9 to 24.3]
  Platelet Response | 0 | 0.0 [0.0 to 10.6]
  Neutrophil Response | 0 | 0.0 [0.0 to 10.6]

8. Secondary Outcome: Percentage of Participants With Complete Remission (CR) and Marrow CR
Description: Percentage of participants with CR and marrow CR were reported. CR per International Working Group (IWG) 2006 Response criteria: Bone marrow - less than or equal to (<=)5% myeloblasts with normal maturation of all cell lines, persistent dysplasia noted; Peripheral blood - hemoglobin >=11 g/dL; platelets >=100*10^9/L; neutrophils >=1.0*10^9/L; blasts, 0%. Marrow CR: Bone marrow - <=5% myeloblasts and decrease by >=50% over pretreatment; Peripheral blood - if HI responses, they were noted in addition to marrow CR.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants
  Complete Remission (CR) | 0 | 0
  Marrow CR | 0 | 3.0

9. Secondary Outcome: Percentage of Participants With Partial Remission (PR)
Description: Percentage of participants with PR were reported. PR per International Working Group (IWG) 2006 Response criteria: All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by >=50% over pretreatment but still >5%, cellularity and morphology not relevant.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants With Cytogenetic Response
Description: Percentage of participants with cytogenetic response were reported. Cytogenetic response per International Working Group (IWG) 2006 Response criteria: Complete - disappearance of the chromosomal abnormality without appearance of new ones; Partial - at least 50% reduction of the chromosomal abnormality.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Percentage of participants | 0 | 0

11. Secondary Outcome: Overall Survival
Description: The overall survival was defined as the time from the date of first dose of study drug to date of death from any cause. Median overall survival was estimated by using the Kaplan-Meier method.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Months | NA [NA to NA] — Here, NA signifies that the median, lower and upper limit of Confidence Interval (CI) could not be calculated for single participant. | NA [NA to NA] — Here, NA signifies that the median, lower and upper limit of Confidence Interval (CI) were not estimable due to lesser number of events.

12. Secondary Outcome: Time to Progression to Acute Myeloid Leukemia (AML)
Description: Time to progression to acute myeloid leukemia was reported. Disease progression as per IWG response criteria: For participants with:
  <5% blasts: >=50% increase in blasts to >5% blasts; 5%-10% blasts: >=50% increase to >10% blasts; 10%-20% blasts: >=50% increase to >20% blasts; 20%-30% blasts: >=50% increase to >30% blasts. Any of the following: >=50% decrement from maximum remission/response in granulocytes or platelets; reduction in hemoglobin by >=2 g/dL; transfusion dependence.
Time Frame: Up to 2 years
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Talacotuzumab | Daratumumab
Number analyzed (Participants) | 1 | 33
Weeks | NA [NA to NA] — Here, NA signifies that the median, lower and upper limit of Confidence Interval (CI) could not be calculated for single participant. | NA [54.7 to NA] — Here, NA signifies that the median and upper limit of Confidence Interval (CI) were not estimable due to lesser number of events.

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Talacotuzumab | Daratumumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 6/33
Serious Adverse Events (participants affected / at risk) | 1/1 | 15/33
Other Adverse Events (participants affected / at risk) | 1/1 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talacotuzumab (N=1) | Daratumumab (N=33)
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Autoimmune Disorder (Immune system disorders) | 0 | 1
Corona Virus Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Lung Infection Pseudomonal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talacotuzumab (N=1) | Daratumumab (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9
Atrial Fibrillation (Cardiac disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Conjunctival Haemorrhage (Eye disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 7
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 0 | 6
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 6
Oedema Peripheral (General disorders) | 0 | 6
Peripheral Swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 3
Campylobacter Infection (Infections and infestations) | 0 | 2
Herpes Simplex (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 3
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 4
Blood Creatinine Increased (Investigations) | 0 | 2
Weight Decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 0 | 5
Paraesthesia (Nervous system disorders) | 0 | 2
Renal Impairment (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 5
Hypotension (Vascular disorders) | 0 | 2
Pallor (Vascular disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study objectives were not pursued in talacotuzumab arm; enrollment in this arm was stopped due to a serious infusion-related reaction after first dose in first participant assigned to talacotuzumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT03011034/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT03011034/SAP_001.pdf